CLINICAL TRIAL: NCT00578097
Title: A Phase II, International, Multi-centre, Prospective, Randomised, Parallel-group, Double-blind, Dose-ranging, Placebo-controlled, 12-week, Princeps Study to Assess the Efficacy and Safety of a One Injection Cycle With Either Botulinum Toxin Type-A (Dysport® 125, 250 or 500 Units) or Placebo Followed by an Optional 6-month Extension Phase in the Symptomatic Treatment of Micturition Urgency and Frequency in Continent Female Subjects Suffering From Idiopathic Overactive Bladder.
Brief Title: Efficacy and Safety Study of Botulinum Toxin Type-A (Dysport®) in Continent Female Subjects Suffering From Idiopathic Overactive Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to poor recruitment.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-79-52120-126; 2007-002999-34 (EudraCT Number)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A - 125 units (Experimental)
  Interventions: Biological: Botulinum toxin type A
- B - 250 units (Experimental)
  Interventions: Biological: Botulinum toxin type A
- C - 500 units (Experimental)
  Interventions: Biological: Botulinum toxin type A
- D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — Single injection cycle, intradetrusor injection at baseline visit 2 of either 125 units (arm A), 250 units (arm B) or 500 units (arm C) in total.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: A - 125 units; B - 250 units; C - 500 units
Drug: Placebo — Single injection cycle, intradetrusor injection at baseline (visit 2).
  Arms: D

SUMMARY:
The purpose of this study is to determine the optimal dose of botulinum toxin type A injected in the detrusor muscle to improve urinary symptoms, urodynamic parameters and quality of life of continent women suffering from idiopathic overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a diagnosis of idiopathic overactive bladder, without incontinence.
* The subject has ≥ 3 urgency episodes over the course of the 3 days immediately preceding the Baseline visit.
* The subject has ≥ 24 episodes of micturition over the course of the 3 days immediately preceding the Baseline visit.

Exclusion Criteria:

* Bladder outlet obstruction (on urodynamic assessment).
* Post-Micturition Residual Volume > 150 ml (ultrasound assessment).
* Evidence of a urinary tract infection at Screening or Baseline in the study.
* Active or history of interstitial cystitis, malignancy of the bladder or urothelial tract, a carcinoma in situ (non malignant melanoma is allowed) bladder and/or kidney stones.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of episodes of urgency and frequency of micturition. | Week 12

SECONDARY OUTCOMES:
The number of episodes of urgency, frequency of micturition, and frequency of nocturia. | All timepoints
Severity of urgency. | All timepoints
Maximum flow rate and post-micturition residual volume (PMRV). | Day 4 and Week 6
Standard International Continence Society (ICS) urodynamic parameters. | Week 12
Quality of Life (QoL). | All timepoints
Safety | All timepoints
Extension study - Duration of effect as determined by the persistence of a positive response. | All timepoints
Extension study - The number of episodes of urgency, frequency of micturition, and frequency of nocturia. | All timepoints
Extension study - Severity of urgency. | All timepoints
Extension study Quality of Life (QoL) | All timepoints
Extension study safety. | All timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (34):
- Belgium (4):
  - ULB Hôpital Erasme, Brussels
  - CH Régional Huy - Polyclinique A Rue Trois Ponts, Huy
  - UZ Gasthuisberg, Leuven
  - CHU Liege Sart Tilman, Liège
- Czechia (2):
  - Urologická klinika, Olomouc
  - Urologické oddělení, Prague
- France (5):
  - Hôpital Michallon - CHU de Grenoble, Grenoble
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Hôpital Charles Nicolle - CHU de Rouen, Rouen
  - Hôpital Henri Gabrielle - Hôpitaux Civils de Lyon, Saint-Genis-Laval
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
- Germany (8):
  - Medizinische Einrichtungen der RWTH, Aachen
  - Praxis für Urologie, Bad Kreuznach
  - Praxis für Urologie, Emmendingen
  - Praxis für Urologie, Günzburg
  - Praxis für Urologie, Lahr
  - Beckenboden Zentrum München, München
  - Städtisches Klinikum Neunkirchen gGmbH, Neunkirchen
  - Krankenhaus St. Trudpert, Pforzheim
- Italy (3):
  - Unità Spinale, Azienda Ospedaliera Careggi, Florence
  - Unità Spinale, Ospedale Niguarda, Milan
  - Struttura Complessa di Neuro-Urologia, Torino
- Netherlands (4):
  - General Urology Academisch Ziekenhuis Maastricht, Maastricht, P.Debyelaan 25
  - VU Medisch Centrum Amsterdam, Amsterdam
  - UMC St. Radboud, Nijmegen
  - Erasmus MC, Universitair Medisch Centrum Rotterdam, Rotterdam
- Spain (3):
  - Hospital San Rafael, Madrid
  - Hospital Clínico Universitario Canarias, San Cristóbal de La Laguna
  - Hospital Universitario La Fe, Valencia
- United Kingdom (5):
  - Southmead Hospital, Bristol
  - Western General Hospital, Edinburgh
  - St George's Hospital, London
  - Churchill Hospital, Oxford
  - Royal Berkshire Hospital, Reading